CLINICAL TRIAL: NCT02532114
Title: A Phase I Study of Niclosamide in Combination With Enzalutamide in Men With Castration-Resistant Prostate Cancer
Brief Title: Niclosamide and Enzalutamide in Treating Patients With Castration-Resistant, Metastatic Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9390; NCI-2015-01246 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CC9390; 9390 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); P50CA097186 (NIH)
Record Dates: First submitted 2015-08-12; First posted 2015-08-25 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Castration Levels of Testosterone; Castration-Resistant Prostate Carcinoma; Metastatic Prostate Carcinoma; Recurrent Prostate Carcinoma; Stage IV Prostate Adenocarcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; Niclosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (niclosamide, enzalutamide) (Experimental): Patients receive niclosamide PO TID and enzalutamide PO daily. Treatment continues for 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Enzalutamide; Other: Laboratory Biomarker Analysis; Drug: Niclosamide; Other: Pharmacological Study

INTERVENTIONS:
Drug: Enzalutamide — Given PO
  Other Names: ASP9785; MDV3100; Xtandi
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Niclosamide — Given PO
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of niclosamide when given together with enzalutamide in treating patients with castration resistant prostate cancer that has spread from the primary site to other places in the body. Androgens such as testosterone can cause the growth of prostate cancer cells. Drugs like enzalutamide block androgens from driving tumor growth; however, when androgen receptor splice variants are present, these drugs may not be effective. Niclosamide may decrease the amount of androgen receptor splice variant present within tumor cells, thus promoting the anti-tumor effects of enzalutamide. Giving niclosamide together with enzalutamide may be a better treatment for prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and tolerability of three-times-daily (TID) oral niclosamide combined with enzalutamide in men with castration-resistant prostate cancer (CRPC) that has progressed on abiraterone (abiraterone acetate).

SECONDARY OBJECTIVES:

I. Determine the effect of niclosamide plus enzalutamide on androgen receptor splice variant (AR-V) expression as determined by quantitative reverse-transcriptase-polymerase-chain-reaction (qRT-PCR).

II. Determine the pharmacokinetic profile of three-times-daily (TID) oral niclosamide in men with castration-resistant prostate cancer (CRPC) that has progressed on abiraterone.

III. Determine the prostate specific antigen (PSA) response rate (i.e. proportion of subjects with >= 50% decline in PSA from pre-study baseline) after 28-days of niclosamide plus enzalutamide.

IV. Determine the effect of niclosamide plus enzalutamide on protein expression and the transcriptional program of circulating tumor cells.

OUTLINE: This is a dose-escalation study of niclosamide.

Patients receive niclosamide orally (PO) TID and enzalutamide PO daily. Treatment continues for 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at days 58 and 88.

ELIGIBILITY:
Inclusion Criteria:

* Have signed an informed consent document indicating that the subject understands the purpose of and procedures required for the study and are willing to participate in the study
* Be willing/able to adhere to the prohibitions and restrictions specified in this protocol
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Documented histologically confirmed adenocarcinoma of the prostate
* Patient must have evidence of castration resistant prostate cancer as evidenced by a confirmed rising PSA (per Prostate Cancer Working Group 2 [PCWG2] criteria) and a castrate serum testosterone level (i.e. =< 50 mg/dL)
* Patient must be eligible for treatment with enzalutamide
* Patient must have previously progressed on abiraterone (either by PCWG2 criteria or Response Evaluation Criteria in Solid Tumors [RECIST] criteria)
* Documented metastatic disease on bone scan, computed tomography (CT) scan or magnetic resonance imaging (MRI)

Exclusion Criteria:

* Have known allergies, hypersensitivity, or intolerance to enzalutamide or niclosamide or their excipients
* Ongoing systemic therapy (other than a gonadotropin releasing hormone [GnRH] agonist/antagonist) for prostate cancer including, but not limited to:

  * Cytochrome P450, family 17 (CYP-17) inhibitors (e.g. ketoconazole, abiraterone)
  * Antiandrogens (e.g. bicalutamide, nilutamide)
  * Second generation antiandrogens (e.g. ARN-509)

    * Note: patients receiving ongoing treatment with enzalutamide will be allowed to join the study
  * Immunotherapy (e.g. sipuleucel-T, ipilimumab)
  * Chemotherapy (e.g. docetaxel, cabazitaxel)
  * Radiopharmaceutical therapy (e.g. radium-223, strontium-89, samarium-153)
* Have any condition that, in the opinion of the investigator, would compromise the well-being of the subject or the study or prevent the subject from meeting or performing study requirements
* Any psychological, familial, sociological, or geographical condition that could potentially interfere with compliance with the study protocol and follow-up schedule
* Severe hepatic impairment (Child-Pugh class C)
* Severe renal impairment (creatinine clearance =< 30 ml/min)
* History of prior seizures
* Central nervous system metastases
* Symptomatic patients who, in the opinion of the investigator, may benefit from docetaxel-based chemotherapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-12-31 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities, graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 28 days
Recommended phase 2 dose | Up to 28 days

SECONDARY OUTCOMES:
Half-life of niclosamide | 0.5, 1, 1.5, 2, 3, 4, 6, and 8 hours and 15 days after the first dose of niclosamide
  Mean niclosamide concentration versus time will be plotted for each dose cohort. Half-life will be reported as a mean for each dose cohort along with the observed ranges.
Maximum concentration of niclosamide | 0.5, 1, 1.5, 2, 3, 4, 6, and 8 hours and 15 days after the first dose of niclosamide
  Mean niclosamide concentration versus time will be plotted for each dose cohort. maximum concentration will be reported as a mean for each dose cohort along with the observed ranges.
Minimum concentration of niclosamide | 0.5, 1, 1.5, 2, 3, 4, 6, and 8 hours and 15 days after the first dose of niclosamide
  Mean niclosamide concentration versus time will be plotted for each dose cohort. Minimum concentration will be reported as a mean for each dose cohort along with the observed ranges.
PSA response rate | Baseline to up to 28 days
  The percent change in PSA will be presented as a waterfall plot, with the rate of PSA response (i.e. >= 50% decline in PSA from baseline) reported as percentages with 95% confidence intervals.
Steady state concentration of niclosamide | 0.5, 1, 1.5, 2, 3, 4, 6, and 8 hours and 15 days after the first dose of niclosamide
  Mean niclosamide concentration versus time will be plotted for each dose cohort. Steady state concentration will be reported as means for each dose cohort along with the observed ranges.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schweizer, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Schweizer MT, Haugk K, McKiernan JS, Gulati R, Cheng HH, Maes JL, Dumpit RF, Nelson PS, Montgomery B, McCune JS, Plymate SR, Yu EY. A phase I study of niclosamide in combination with enzalutamide in men with castration-resistant prostate cancer. PLoS One. 2018 Jun 1;13(6):e0198389. doi: 10.1371/journal.pone.0198389. eCollection 2018. PMID 29856824